CLINICAL TRIAL: NCT05977777
Title: Characterization of Pancreatic Lesions Using Dynamic Contrast-enhanced Ultrasound
Brief Title: Contrast-enhanced Ultrasound and Pancreatic Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Zocco Maria Assunta, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5220
Record Dates: First submitted 2023-03-16; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients affected by focal pancreatic lesions
  Interventions: Diagnostic Test: Contrast- enhanced ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast- enhanced ultrasound — Contrast- enahnched ultrasound is performed on target pancreatic lesion

SUMMARY:
The characterization of pancreatic lesions is one of the fundamental steps in the management of pancreatic neoplastic diseases. In terms of a subjective assessment of vascular enhancement in the various examination stages, the use of contrast-enhanced ultrasonography (CEUS) in the study of pancreatic neoplastic disease has been thoroughly investigated. Technology advancements have enabled the development of software that can perform an objective study of the parameters of vascular enhancement and their variations during dynamic CEUS (DCEUS). Currently, the paucity of data regarding the characterization of pancreatic lesions trough DCEUS limit the definition of its role in pancreatic disease. The main purpose of this study is to employ the knowledge in this field trough the characterization of focal pancreatic lesions using DCEUS.

DETAILED DESCRIPTION:
Pancreatic cancer is currently one of the most prevalent malignant neoplasms, characterized by an increasing prevalence and a high mortality and lethality rate. It is the seventh most common malignant tumor in the general population, the fourth most deadly in both sexes, with a 5-year survival rate of approximately 9%. The lack of an early diagnostic tool and the absence of effective treatments for advanced-stage disease are the major contributors to this poor prognosis.

The diagnosis of pancreatic cancer is based on the results of multiple examinations, including various imaging modalities, until the histological diagnosis is obtained through biopsy. Transabdominal ultrasound (US) computed tomography (CT), magnetic resonance imaging (MRI), and endoscopic ultrasound (EUS) are performed to detect and stage pancreas cancer in resectable, borderline, locally advanced and metastatic. Hence, the differential diagnosis and characterization of solid pancreatic tumors represent a crucial step in identifying a suitable therapeutic strategy.

Transabdominal US is frequently used as a first-line diagnostic tool for patients with suspected pancreatic diseases. The main limitation of transabdominal US is the low accuracy in the differential diagnosis between malignant and benign solid lesions, and, considering malignant lesions, between the different pancreatic tumors (adenocarcinomas, neuroendocrine tumors, carcinosarcomas, lymphomas) since all these masses appear as hypoechoic formations.

The introduction of ultrasound contrast agent (UCA) has significantly improved the diagnostic abilities of conventional ultrasound and contrast enhanced ultrasound (CEUS) has been widely implemented in clinical practice because of the enormous quantity of information it provides, along with its low cost, reproducibility, minimal invasiveness, and safety of the UCA. In the detection of pancreatic cancer, contrast enhanced ultrasound (CEUS) achieve a sensitivity and specificity of 92% and 76%, respectively. The European Federation for Ultrasound in Medicine and Biology (EFSUMB) has recently defined the importance of contrast-enhanced ultrasonography (CEUS) in the diagnosis of pancreatic disease, supporting its use to characterize B-mode-identified pancreatic solid lesions.

Despite its numerous advantages, one of the most significant limitations of CEUS is the subjective evaluation of contrast enhancement related behavior of tissues examined. In recent years, one of the methods explored to overcome this limitation has been the Dynamic CEUS (DCEUS) which allow the quantitative analysis of UCA-kinetics in a specific region of interest (ROI). It consists of measuring the average intensity of a ROI following a bolus injection of UCA and generating a time-intensity curve (TIC). Then, multiple parameters are derived from the TIC to quantitatively characterize the different stages of the wash-in and wash-out phases. These parameters can be divided into three categories: time parameters, intensity parameters and area under the curve (AUC).

Very few evidence has been published concerning the use of DCEUS in the characterization of pancreatic lesions. Kersting et al performed DCEUS in sixty undetermined pancreatic lesions then histologically characterized as pancreatic ductal adenocarcinoma (PDAC) (n = 45) or inflammatory lesion in chronic pancreatitis (CP) (n = 15). The grouped analysis of TICs showed a significant prolonged time to peak and arrival time for PDAC then CP compared with normal pancreatic tissue. In another study, D'Onofrio et al performed a quantitative perfusion analysis of ten prospectively enrolled patients with suspected pancreatic ductal adenocarcinoma (PDAC). The results showed a significant difference in peak of enhancement and ascending curve between PDAC and normal pancreatic parenchyma, providing an objective quantification of enhancement for the assessment of pancreatic lesion. These findings suggest a potential usefulness of DCEUS in characterizing and differentiating focal pancreatic lesions. However, the amount of data currently available in the published studies is limited.

The main purpose of this study is to employ the knowledge in this field trough the characterization of focal pancreatic lesions using DCEUS.

Materials and methods Fifty patients with a transabdominal US diagnosis of a pancreatic lesion who receive CEUS and a subsequent biopsy for histologic characterization will be enrolled in this prospective study. Inclusion criteria are at least 18 years of age, at least one pancreatic lesion visible in B-mode US and investigated trough CEUS and provide written consent. Exclusion criteria comprise less than 18 years of age and absence of informed consent.

All patients enrolled in this study will be fasting for at least 8 hours before CEUS examinations. During the B-mode ultrasound, location, size and echogenicity of lesion detected will be assess. According to CEUS guideline, after the bolus injection of 2.4 ml sulfur hexafluoride microbubbles (SonoVue/Lumason, Bracco) via peripheral upper limb vein and followed by a 5-10 ml saline flush, the enhancement features of the lesion during arterial, portal, and late phases will be recorded and examined. Clinical and laboratoristic data will be also recorded. After examination, TICs will be obtained and the following quantitative parameters will be described: peak enhancement, time to peak, area under the curve, mean transit time and the slope of wash-in curve.

Statistical analysis This is monocenter, prospective, non-pharmacological trial. Nominal or ordinal variables will be presented as frequencies and percentages. Mean, standard deviation, median and 95% confidence intervals will be calculated for continuous variables. Comparison between means/median will be investigated with Mann-Whitney test. A p value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria are:

* written informed consent
* at least 18 years of age
* at least one pancreatic lesion visible in B-mode US and investigated trough CEUS

Exclusion criteria:

* less than 18 years of age
* absence of informed consent
* knowm allergy to ultrasound contrast agent
* hearth failure
* pregnancy
* lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
diagnostic agreement between contrast-enhanced ultrasound and histology | within 3 months from enrollement
  to quantify peak enhancement intensity in Arbitray Units AU (measured by analysing D-CEUS time-intensity curves) in patients with pancreatic lesions, stratified according to the histologic exam of pancreatic lesions

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy